CLINICAL TRIAL: NCT00046852
Title: High-Dose Therapy and Autologous Blood Stem Cell Transplantation (ASCT) Followed by Post-Transplant Immunotherapy With Costimulated Autologous T-Cells in Conjunction With Pneumococcal Conjugate Vaccine Immunization for Patients With Multiple Myeloma
Brief Title: Chemotherapy and Peripheral Stem Cell Transplantation Followed By Immunotherapy in Treating Patients With Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: University of Maryland Greenebaum Cancer Center (Other)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000256870; MSGCC-0065; UPCC-6401; NCI-V02-1709
Record Dates: First submitted 2002-10-03; First posted 2003-01-27 (Estimated); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Infection; Multiple Myeloma and Plasma Cell Neoplasm
Keywords: infection; refractory multiple myeloma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Infections; Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Filgrastim; Pneumococcal Vaccines; Carmustine; Cyclophosphamide; Melphalan; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: filgrastim
Biological: pneumococcal polyvalent vaccine
Biological: therapeutic autologous lymphocytes
Biological: therapeutic tumor infiltrating lymphocytes
Drug: carmustine
Drug: cyclophosphamide
Drug: melphalan
Procedure: bone marrow ablation with stem cell support
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining chemotherapy with autologous peripheral stem cell transplantation and immunotherapy may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells. Biological therapies use different ways to stimulate the immune system and stop cancer cells from growing.

PURPOSE: Randomized phase I/II trial to study the effectiveness of combining chemotherapy with peripheral stem cell transplantation followed by immunotherapy in treating patients who have multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of expanding ex vivo autologous T cells and infusing these cells after high-dose chemotherapy and autologous peripheral blood stem cell rescue in patients with multiple myeloma.
* Determine the response rate and progression-free survival of patients who receive anti-CD3/anti-CD28 expanded autologous T cells on either day 14 or day 100 post-transplantation.
* Compare response and survival rates of these patients to historical controls.
* Determine the optimal schedule for pneumococcal conjugate vaccine (PCV) to induce an anti-pneumococcal immune response post-transplantation in these patients.
* Determine whether "vaccine education" of antigen-presenting cells (APCs) in the stem cell graft results in an earlier and/or enhanced immune response than with a graft containing "non-educated" APCs in these patients.
* Determine whether an infusion of T cells presensitized to the PCV and expanded ex vivo contributes to the anti-pneumococcal immune response in these patients.

OUTLINE: This is a randomized, multicenter study.

Patients receive cyclophosphamide IV over 12 hours on day 1 and filgrastim (G-CSF) subcutaneously (SC) daily beginning on day 2. Patients undergo leukapheresis to collect mononuclear cells for autologous T cells (ATCs) and peripheral blood stem cells (PBSCs). ATCs are generated by ex vivo expansion for 8-14 days and selection for CD3+/CD28+ cells.

Patients then receive high-dose therapy comprising carmustine IV over 2 hours on day -2 and melphalan IV over 20 minutes on day -1 or melphalan IV alone on days -2 and -1 (or day -1 only). Autologous PBSCs are reinfused on day 0. Patients also receive G-CSF SC beginning on day 1 and continuing until blood counts recover.

Patients who choose to receive pneumococcal conjugate vaccine (PCV) are randomized to 1 of 4 treatment arms.

* Arm I: Patients receive PCV intramuscularly prior to transplantation (10-14 days before lymphocyte collection) and post-transplantation (1 and 3 months) plus costimulated ATCs IV over 20-60 minutes around day 12-14 post-transplantation.
* Arm II: Patients receive PCV as in arm I but receive ATCs around day 100 post-transplantation.
* Arm III: Patients receive PCV post-transplantation only (at 1 and 3 months) plus ATCs as in arm I.
* Arm IV: Patients receive PCV as in arm III and ATCs as in arm II. Patients who choose not to receive the PCV receive ATCs on about day 12-14 after PBSC transplantation.

All patients are offered standard pneumococcal polysaccharide vaccine at 12 months.

Patients are followed twice weekly until day 60, weekly for 4 months, monthly for 6 months, and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 16-46 patients will be accrued for this study within 14 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of multiple myeloma requiring systemic treatment
* No obvious myelodysplastic changes in the marrow

PATIENT CHARACTERISTICS:

Age

* 18 to 80

Performance status

* ECOG 0-2 (ECOG 3-4 allowed if based solely on bone pain)

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* No chronic active hepatitis
* No liver cirrhosis

Renal

* Creatinine no greater than 3.0 mg/dL
* No dialysis

Cardiovascular

* LVEF at least 45% unless no evidence of untreated clinically significant functional impairment

Pulmonary

* FEV_1 and FVC at least 50% of predicted
* Total lung capacity at least 50% of predicted
* DLCO at least 50% of predicted
* Mild to moderate pulmonary impairment (lower DLCO) allowed but patients would not receive study carmustine
* Patients unable to complete pulmonary function test due to bone pain or fracture must have high-resolution CT scan of the chest and arterial partial pressure of oxygen greater than 70

Other

* No active infections requiring IV antibiotics
* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Prior pulse dexamethasone (1-2 courses) allowed
* Concurrent pulse dexamethasone allowed during mobilization therapy

Radiotherapy

* Not specified

Surgery

* Not specified

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-12; Primary Completion 2004-11 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron P. Rapoport, MD, Study Chair — University of Maryland Greenebaum Cancer Center
Locations (2):
- United States (2):
  - Marlene and Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania